CLINICAL TRIAL: NCT02941484
Title: A Prospective, Randomized Trial of Early Oral Intake After Pancreaticoduodenectomy in the Age of ERAS
Brief Title: Early Oral Intake After Pancreaticoduodenectomy in the Age of ERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zheng Chen, the director of general surgery;, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XuzhouMedSch
Record Dates: First submitted 2016-10-16; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Periampullary Carcinoma Resectable; Pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 early oral intake (Experimental): early oral intake since postoperative day 1.
  Interventions: Procedure: early oral intake
- 2 jejunostomy tube feeding (JTF) (Experimental): jejunostomy tube feeding (JTF) was carried out after PD
  Interventions: Procedure: jejunostomy tube feeding (JTF)

INTERVENTIONS:
Procedure: early oral intake — early oral intake is started within 24 hours after pancreaticoduodenectomies following to the ERAS guideline
  Arms: 1 early oral intake
Procedure: jejunostomy tube feeding (JTF) — The jejunostomy tube was placed using the Flocare CH-10 tube with the longitudinal Witzel jejunostomy technique.nutrition is supplemented via JTF rather than early oral intake.Velocity is progressively increased by 20ml/hr until full nutritional goal (25Kcal/Kg)
  Arms: 2 jejunostomy tube feeding (JTF)

SUMMARY:
Early oral intake after Pancreaticoduodenectomy is recommended strongly according to the ERAS guideline, which was based on studies in patients with gastrointestinal cancer, mainly colorectal and gastric. Specific clinical study on early oral intake after PD is very limited. inadequate nutritional intake was significantly associated with a high incidence of postoperative complications. Therefore, the present study is aim to evaluate the tolerance, safety, and efficacy in the patients undergoing PD in the age of ERAS.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery (ERAS) is an interdisciplinary, multimodal concept and has become an important focus of Pancreaticoduodenectomy procedures following universal accepted and practice in gastrointestinal and colorectal surgeries. Early oral diet without restrictions after operation is recommended strongly according to ERAS guideline. However, several studies demonstrated that only half validated the true practice of the postoperative oral diet. Furthermore, Oral intake tolerance after PD is controversial. Only 23% of patients were able to take solid food at day 3. It appears that adequate nutritional intake only via oral diet is a severe challenge. Besides, Studies showed that insufficient amount of dietary intake was significantly associated with extended duration of postoperative hospitalization and parenteral nutrition. Importantly, Specific clinical study on early oral intake after PD is very limited. Therefore, the present study is aim to evaluate the tolerance, safety, and efficacy in the patients undergoing PD in the age of ERAS.

ELIGIBILITY:
Inclusion Criteria:

* Periampullar carcinoma
* Pancreaticoduodenectomy
* ERAS protocol implemented

Exclusion Criteria:

* Preoperative Radiotherapy/chemotherapy
* Unresectable primary cancer
* Palliative surgery
* New York Heart Association class>3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Tolerance of Oral Intake | postoperative 1 to 7day
  the amount of oral intake is recorded, including clear fluids, soft and solid food.

SECONDARY OUTCOMES:
morbidity rate | postoperative 1day to discharge, up to 8 weeks
  complications associated with surgery, early oral intake,and jejunostomy tube.Definitions used for specific complications are according to the International Study Group on Pancreatic Fistula (ISGPF) definition.
length of stay | postoperative 1day to discharge,up to 8 weeks
  postoperative length of stay
Readmission rate | 30 days after discharge
Hospital costs | postoperative 1day to discharge,up to 8 weeks
Albumin | postoperative 30d
  serum albumin
weight | postoperative 30d
  weight in kilograms
height | postoperative 30d
  height in meters

CONTACTS AND LOCATIONS:
Overall Officials: zheng chen, MD;PHD, Principal Investigator — Xuzhou Medical University Affiliated Suqian Hospital
Locations (1):
- Suqian Hospital, Suqian, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bozzetti F, Mariani L. Perioperative nutritional support of patients undergoing pancreatic surgery in the age of ERAS. Nutrition. 2014 Nov-Dec;30(11-12):1267-71. doi: 10.1016/j.nut.2014.03.002. Epub 2014 Mar 14. PMID 24973198
- [Background] Buscemi S, Damiano G, Palumbo VD, Spinelli G, Ficarella S, Lo Monte G, Marrazzo A, Lo Monte AI. Enteral nutrition in pancreaticoduodenectomy: a literature review. Nutrients. 2015 Apr 30;7(5):3154-65. doi: 10.3390/nu7053154. PMID 25942488
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Afaneh C, Gerszberg D, Slattery E, Seres DS, Chabot JA, Kluger MD. Pancreatic cancer surgery and nutrition management: a review of the current literature. Hepatobiliary Surg Nutr. 2015 Feb;4(1):59-71. doi: 10.3978/j.issn.2304-3881.2014.08.07. PMID 25713805
- [Background] Lassen K, Coolsen MM, Slim K, Carli F, de Aguilar-Nascimento JE, Schafer M, Parks RW, Fearon KC, Lobo DN, Demartines N, Braga M, Ljungqvist O, Dejong CH; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care for pancreaticoduodenectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. World J Surg. 2013 Feb;37(2):240-58. doi: 10.1007/s00268-012-1771-1. No abstract available. PMID 22956014
- [Background] Nussbaum DP, Penne K, Stinnett SS, Speicher PJ, Cocieru A, Blazer DG 3rd, Zani S, Clary BM, Tyler DS, White RR. A standardized care plan is associated with shorter hospital length of stay in patients undergoing pancreaticoduodenectomy. J Surg Res. 2015 Jan;193(1):237-45. doi: 10.1016/j.jss.2014.06.036. Epub 2014 Jun 26. PMID 25062813
- [Background] Wei J, Chen W, Zhu M, Cao W, Wang X, Shi H, Dong B, Sun J, Chen H, Zhou Y, Zhou S, Xu J; Chinese Medical Association's Nutrition Support Group for Geriatric Patients. Guidelines for parenteral and enteral nutrition support in geriatric patients in China. Asia Pac J Clin Nutr. 2015;24(2):336-46. doi: 10.6133/apjcn.2015.24.2.11. PMID 26078252
- [Background] Weimann A, Braga M, Harsanyi L, Laviano A, Ljungqvist O, Soeters P; DGEM (German Society for Nutritional Medicine); Jauch KW, Kemen M, Hiesmayr JM, Horbach T, Kuse ER, Vestweber KH; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Surgery including organ transplantation. Clin Nutr. 2006 Apr;25(2):224-44. doi: 10.1016/j.clnu.2006.01.015. Epub 2006 May 15. PMID 16698152
- [Background] Bounoure L, Gomes F, Stanga Z, Keller U, Meier R, Ballmer P, Fehr R, Mueller B, Genton L, Bertrand PC, Norman K, Henzen C, Laviano A, Bischoff S, Schneider SM, Kondrup J, Schuetz P; Members of the Working Group. Detection and treatment of medical inpatients with or at-risk of malnutrition: Suggested procedures based on validated guidelines. Nutrition. 2016 Jul-Aug;32(7-8):790-8. doi: 10.1016/j.nut.2016.01.019. Epub 2016 Feb 18. PMID 27160498
- [Background] Joliat GR, Labgaa I, Petermann D, Hubner M, Griesser AC, Demartines N, Schafer M. Cost-benefit analysis of an enhanced recovery protocol for pancreaticoduodenectomy. Br J Surg. 2015 Dec;102(13):1676-83. doi: 10.1002/bjs.9957. Epub 2015 Oct 22. PMID 26492489
- [Background] Coolsen MM, Bakens M, van Dam RM, Olde Damink SW, Dejong CH. Implementing an enhanced recovery program after pancreaticoduodenectomy in elderly patients: is it feasible? World J Surg. 2015 Jan;39(1):251-8. doi: 10.1007/s00268-014-2782-x. PMID 25212064
- [Background] Chaudhary A, Barreto SG, Talole SD, Singh A, Perwaiz A, Singh T. Early discharge after pancreatoduodenectomy: what helps and what prevents? Pancreas. 2015 Mar;44(2):273-8. doi: 10.1097/MPA.0000000000000254. PMID 25479587
- [Background] Bischoff SC, Singer P, Koller M, Barazzoni R, Cederholm T, van Gossum A. Standard operating procedures for ESPEN guidelines and consensus papers. Clin Nutr. 2015 Dec;34(6):1043-51. doi: 10.1016/j.clnu.2015.07.008. Epub 2015 Jul 16. PMID 26254807
- [Background] Braga M, Pecorelli N, Ariotti R, Capretti G, Greco M, Balzano G, Castoldi R, Beretta L. Enhanced recovery after surgery pathway in patients undergoing pancreaticoduodenectomy. World J Surg. 2014 Nov;38(11):2960-6. doi: 10.1007/s00268-014-2653-5. PMID 24870390
- [Background] Coolsen MM, van Dam RM, van der Wilt AA, Slim K, Lassen K, Dejong CH. Systematic review and meta-analysis of enhanced recovery after pancreatic surgery with particular emphasis on pancreaticoduodenectomies. World J Surg. 2013 Aug;37(8):1909-18. doi: 10.1007/s00268-013-2044-3. PMID 23568250